CLINICAL TRIAL: NCT01599403
Title: Comparative Effectiveness of Continuous Thoracic Paravertebral Blocks Versus Thoracic Epidural and Continuous Intercostal Blocks Versus Patient-Controlled Anesthesia in Traumatic Rib Fracture Patients
Brief Title: Thoracic Blocks Versus Thoracic Epidural and Patient Controlled Anesthesia in Traumatic Rib Fracture Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Gyorgy Frendl, Director, Surgical ICU Translational Research (STAR) Center, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2011P002702 Frendl
Record Dates: First submitted 2012-02-28; First posted 2012-05-16 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Traumatic Rib Fracture
Keywords: Rib Fracture; Intercostal Nerve Block; Paravertebral Nerve Block
MeSH Terms: conditions — Rib Fractures | interventions — Anesthesia, Epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Paravertebral Block (Active Comparator): Patients will receive 1 or 2 paravertebral catheters for ongoing infusion of local anesthestic
  Interventions: Procedure: Paravertebral Block
- Patient Controlled Anesthesia (No Intervention): Standard usual care
- Epidural Block (Experimental): Intervention:
  Patients will have epidural catheters placed for the infusion of local anesthetic solution to control pain (if qualified for this approach and randomized here)
  Interventions: Procedure: Epidural Block
- Intercostal Nerve Block (Active Comparator): Patients will receive intercostal catheters for the infusion of local anesthetic solution to control pain(if qualified for this arm and randomized here)
  Interventions: Procedure: Intercostal Nerve Block

INTERVENTIONS:
Procedure: Paravertebral Block — The paravertebral block consists of injection of local anesthetics into the area next to the spinal column and results in regional pain control. This technique of this block may be performed on multiple levels if there are extensive rib fractures and may be performed on both sides of the rib cage depending on injury.
  Arms: Paravertebral Block
Procedure: Intercostal Nerve Block — The intercostal nerve block will consist of placing a catheter which delivers pain medication into the area between the ribs. This technique of this block may be performed on multiple levels if there are extensive rib fractures and may be performed on both sides of the rib cage depending on injury.
  Arms: Intercostal Nerve Block
Procedure: Epidural Block — The epidural block consists of continuous infusion of local anesthetics into the epidural catheter placed into the epidural space (next to the spinal column) and results in regional pain control. This technique of this block may be performed at the appropriate level so the pain of rib fracture may be better controlled.
  Arms: Epidural Block

SUMMARY:
The primary objective of this study is to investigate whether continuous PVB is equal in efficacy to epidural anesthesia in terms of analgesia in patients with INR lower than 1.2, or is continuous ICNB equal in efficacy to PCA in terms of analgesia, if patients have INRs equal to or greater than 1.2.

DETAILED DESCRIPTION:
Rib fractures are the most common injury sustained following blunt trauma. Ziegler and Agarwal noted that in a population of more than 7000 trauma patients, 10% had fractured ribs. These injuries are normally the hallmark of significant chest trauma; and as the number of fractured ribs increases, there is an exponential increase in morbidity and mortality.

This injury therefore poses a challenging problem from both pulmonary and analgesia standpoints. Significant morbidity is often the result of hypoventilation leading to atelectasis, pneumonia, and respiratory failure. Pain management has been recognized as an important factor in preventing these complications.

Good analgesia may help to improve a patient's respiratory mechanics, leading to a decreased need for mechanical ventilatory support, a shortened hospital stay, and can dramatically alter the course of recovery impacting both morbidity and mortality.

For healthy patients with one to two fractured ribs, systemic analgesics may suffice. For more than three to four fractured ribs, studies and experience have reaffirmed the superior analgesia made possible with continuous thoracic epidural, continuous thoracic paravertebral, and continuous intercostal block, however, a comparative head to head trial comparing the relative merits and disadvantages of each technique has not been undertaken in multiple rib fracture patients. Placing a catheter, which is possible with the use of all three techniques, allows the continuation of analgesia for multiple days with just one block, which is an essential option when treating patients that are likely to need extended analgesia.

All options are not available for all patients, however, as the current American Society of Regional Anesthesiology advises against the performance of epidural or paravertebral blocks in patients with abnormal INR (at the BWH, equal or above 1.2, and/or treatment with other anticoagulants such gpIIb/IIIa inhibitors (heparin and heparin-like medications are usually acceptable within certain dosing time frames).

Rib fractures following trauma are associated with severe postoperative pain and significant morbidity. Atelectasis, pneumonia, pulmonary embolism (PE), and intensive care admission are related to poor analgesia and consequent immobility and splinting during inspiration. With traumatic multiple fractured ribs (MFR), concomitant lung injury is expected. The effect of this injury is exacerbated when the pain of MFR leads to guarding, shallow breaths, and suboptimal chest physiotherapy. Atelectasis, pneumonia, consolidation, and respiratory failure ensue, necessitating or prolonging assisted ventilation and/or oxygenation and increasing morbidity and mortality. Additionally, inadequately treated pain after rib fractures can lead to chronic pain and global deconditioning.

Without the implementation of effective regional and/or neuraxial analgesia, the need for the use of sedative and systemic opioid medications increases, which has the potential to increase the length of stay and increase complications such as delirium, aspiration, decreased mobility with subsequent greater deconditioning and increased risk for embolic events, addiction, and possibly chronic pain. These risks are even higher in older individuals (age > 55), in whom comorbidities and poor respiratory reserves conspire to increase morbidity and mortality, and who are less able to handle and recover from the side effects of sedative and systemic opioid medications. Additionally, trauma patients may also be at higher risk due to multiple, and often confounding, injuries.

Options for analgesia aside from regional blocks include the use of NSAIDs, acetaminophen, opioids, ketamine, and transdermal lidocaine (patch). The short-term disadvantages of NSAID include gastric irritation, platelet inhibition and renal injury. Acetaminophen at high doses is hepatotoxic. Powerful opioids are depressants, suppress cough, increase risk of delirium, and may promote respiratory complications even as they reduce pain. Ketamine causes dissociation and risk of hallucinations, often of an unpleasant nature. Assessment of head and abdominal injuries can be compromised by systemic opioids or ketamine. Of note, none of these medications at well tolerated doses are sufficient to greatly diminish the pain of MFR during chest physiotherapy and coughing, delaying recovery, and none of these treatments can, at well tolerated doses, provide sufficient analgesia without causing significant side effects, even in combination. Lidocaine patches over the fracture sites are ineffective.

Regional/neuraxial blocks provide superior analgesia, the impact of a successful block is immediate and substantial, and, especially regarding elderly, some authorities have categorically stated that most 55-65 year-olds with three or four fractured ribs should receive a regional block. The relative lack of systemic sedation makes it easier to monitor patients with head and abdominal injuries, and the reduced need for systemic medications obviates their inherent concomitant risks.

Though effective, the use of epidural blocks in the intubated and unresponsive patient, especially in the thoracic region, is currently not widely accepted for fear of inadvertent adverse neurologic complications. This said, the incidence of neurological complications associated with patients who cannot respond to incidental injury associated with the placement of epidural anesthesia under general anesthesia, as an example of an unresponsive patient, is not precisely known. Horlocker et al state the "possibility of serious complications may still be as high as 0.08%." Regardless of the exact incidence rate, the prevailing wisdom is that the risk benefit ratio does not support the practice of epidural/deep plexus regional anesthesia in unconscious patients because of the clear association of pain during placement or injection and subsequent injury, which speak to the need for feedback from the patient in preventing injury.

In comparison to epidural analgesia, the major complication of PVB and ICNB is that of pneumothorax with no documented accounts of nerve damage due to the lateral anatomic plane of medication delivery in reference to the central nerve axis. However, in patients with a chest tube this risk is effectively obviated. Moreover, the use of ultrasound, which greatly enhances the ability to avoid of the pleura, further improves the accuracy and safety of these blocks.

Additionally, in view of pain relief methods providing the greatest preservation of pulmonary spirometric function after thoracotomy-related rib trauma, the most effective analgesic method is paravertebral analgesia, with patients having approximately 75% of their preoperative values in the first 48 hours after surgery. Most other techniques e.g. traditional intercostal nerve blocks, epidural local anesthetics or local anesthetic-opiate combinations produce approximately a 55% preservation by 48 hours, with interpleural analgesia being the least effective, with a mean of 35% preservation by 48 hours, less even than TENS or cryoanalgesia. These findings suggest that a thoracic paravertebral block is the best available analgesic method in rib trauma patients: however, the above studies have been performed in the post-surgical setting and not the trauma setting, and concentrated their findings on respiratory parameters, and not pain relief, though the two may be related.

The primary question the investigators wish to answer in this study is whether continuous PVB is equal in efficacy to epidural anesthesia in terms of analgesia in patients with INR lower than 1.2, or is continuous ICNB equal in efficacy to PCA in terms of analgesia, if patients have INRs equal to or greater than 1.2 as measured by difference in visual analog pain scores after 48 hours. Secondary questions are: do PVBs and ICNBs result in a favorable side effect profile, lower complication rate, improved pulmonary mechanics, decreased need for intubation, decreased length of intubation, reduced supplemental oxygenation needs, reduced length of stay, improved speed to work with physical therapy and/or occupational therapy, lesser need for short/long term rehabilitation at discharge, and lesser development of chronic pain when compared to epidural block and opioid PCA in rib fracture patients.

ELIGIBILITY:
Eligibility Criteria

A subject must meet the following criteria to take part in the study:

Inclusion Criteria

* Subjects 18 years of age and greater
* Inpatient on the BWH SICU, MICU, or hospital floor ward
* Non-intubated at the time of block placement
* Traumatic Rib Fractures three or greater
* Block able to be placed within 12-24 hours of presentation to the emergency room
* Ability to provide written informed consent.
* Compliance with all ASRA and BWH Regional Anesthesia in Anticoagulated Patient guidelines for coagulation status.

Exclusion Criteria:

* Subject is pregnant
* Subject not expected to survive 48 hours due to traumatic injuries
* Allergy to Ropivacaine or other local anesthetic
* Any significant concomitant injuries potentially confounding data acquisition (e.g., traumatic brain injury, long bone fractures, intra-abdominal injuries)
* Known allergy to lidocaine
* Inability to provide written, informed consent
* Known opioid medication dependence
* Non-compliance with ARSA and BWH Regional Anesthesia in Anticoagulated Patient Guidelines.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Primary Outcome: Difference in Pain Scores at 48hrs | 2 days
  The primary question investigators wish to answer in this study is whether continuous PVB is equal in efficacy to epidural anesthesia in terms of analgesia in patients with INR lower than 1.2, or is continuous ICNB equal in efficacy to PCA in terms of analgesia, if patients have INRs equal to or greater than 1.2 as measured by visual analog pain scales at 48 hours post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Gyorgy Frendl, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States